CLINICAL TRIAL: NCT02509195
Title: An Open Label Study to Investigate the Safety and Efficacy of Abacavir/Lamivudine/Dolutegravir and the Pharmacokinetic Profile of Dolutegravir in HIV-infected Patients of 60 Years of Age and Older
Brief Title: SSAT064: Pharmacokinetics of Abacavir/Lamivudine/Dolutegravir in HIV Patients of 60 Years and Over
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: St Stephens Aids Trust (Other)
Collaborators: ViiV Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SSAT064; 2014-004970-40 (EudraCT Number)
Record Dates: First submitted 2015-07-08; First posted 2015-07-27 (Estimated); Last update posted 2018-02-28 (Actual); Status verified 2018-02

CONDITIONS: HIV
MeSH Terms: interventions — abacavir, dolutegravir, and lamivudine drug combination

ARMS (1):
- Switch to Triumeq (Experimental): HIV-1 infected subjects currently receiving stable antiretroviral therapy switch their treatment to abacavir/lamivudine/dolutegravir (Triumeq).
  Interventions: Drug: Triumeq

INTERVENTIONS:
Drug: Triumeq — Subjects will take the last dose of their current antiretroviral combination at its usual time on the day before the baseline visit (day 1) and will switch on day 1 to Abacavir/lamivudine/dolutegravir 600mg/300mg/50mg (Triumeq) fixed dose combination once daily between day 1 and day 180.
  Other Names: abacavir/lamivudine/dolutegravir

SUMMARY:
The purpose of this study is to identify the effects that ageing may have on the drug levels, the safety and the efficacy of Dolutegravir.

These effects will be measured in people who are aged 60 or over and taking antiretroviral therapy for HIV infection.

Dolutegravir is a newly licenced anti HIV medication, which belongs to a class of drugs called Integrase Inhibitors. It is taken with two other wellknown agents, Abacavir and Lamivudine, as part of a one tablet once a day regimen, called Triumeq. There is little data available on Dolutegravir in the context of older age. The HIV population is ageing and the investigators know that older age can significantly change the effects and side effects of medications, including that of antiretrovirals.

The investigators aim to investigate the treatment outcomes in older people taking Dolutegravir including the tolerability, efficacy and safety of the drug.

The study will also assess the quality of life (wellbeing of individuals) and cognition (mental abilities) of people aged 60 or over, taking Dolutegravir. The results from this study may inform treatment choices and monitoring in this population in the future.

The duration of involvement in the study will be 6 months with an additional screening visit and a checkup visit 10 days after end of study visit.

DETAILED DESCRIPTION:
Protocol Number: SSAT 064

EudraCT Number: 2014-004970-40

Name of Investigational Product:Triumeq®

Name of active ingredients:Abacavir/lamivudine/dolutegravir

Study title: An open label study to investigate the safety and efficacy of abacavir/lamivudine/dolutegravir and the pharmacokinetic profile of dolutegravir in HIV-infected patients of 60 years of age and older

Objectives:

Primary:

* To assess the steady state pharmacokinetics of dolutegravir 50 mg once daily in HIV-infected subjects of 60 years or greater

Secondary:

* To assess the safety, tolerability, patient quality of life and sleep quality and maintenance of HIV viral load control of abacavir/lamivudine/dolutegravir once daily in HIV-infected subjects of 60 years or greater
* To measure the metabolic profile in patients over the age of 60 with HIV infection who switch antiretroviral regime (metabonomics)
* To investigate cerebral function via cognitive testing before and after a switch in antiretroviral therapy to dolutegravir containing regimens
* To investigate the relationship between genetic polymorphisms and exposure to dolutegravir

Study design:Multi -centre, 180 days (excluding screening and follow up), open label, prospective, one phase pharmacokinetic/pharmacodynamic study

Indication:HIV-1 infection

Methodology:HIV-1 infected subjects will be recruited from four different HIV clinics. Eligible subjects currently receiving stable antiretroviral therapy with an undetectable plasma HIV RNA and with no evidence of previous HIV resistance mutations on genotypic resistance testing, will switch their treatment to abacavir/lamivudine/dolutegravir and undergo a 24 hour pharmacokinetic assessment at day 28 (+/- 1). Monitoring of adverse events (not at screening), viral load, quality of life and sleep quality, will occur at screening and on days 1, 28, 90, and 180. Cognitive function will be tested at screening, baseline and day 180. A sleep diary will be completed between day 1 and day 28.

Planned sample size:A sample size of 40 patients would provide at least 80% power to detect changes in dolutegravir exposure in older people.

Up to 45 subjects may be screened to have 40 patients completing the study.

Summary of eligibility criteria:HIV-1 infected subjects currently receiving stable antiretroviral therapy with undetectable plasma HIV RNA and no evidence of previous HIV- resistance mutations on genotypic resistance testing, 60 years old or older (approximately 30% between 60 and 64 and approximately 70% above the age of 65)

Number of study centres: 4 centres:

Chelsea and Westminster Hospital, London Royal Sussex County Hospital, Brighton St. Mary's Hospital Clinical Trials Centre, London Mortimer Market Centre, UCL, London

Duration of treatment: 180 (+/- 7) days

Dose and route of administration: All study drugs will be administered orally to subjects with the following schedule: Abacavir/lamivudine/dolutegravir one pill once daily

Criteria for evaluation:

Pharmacokinetic parameters of dolutegravir will be evaluated on blood drawn on day 28 (+/- 1) at 0 (pre-dose), 1, 2, 3, 4, 8, 12 and 24 hours post dose.

Monitoring of adverse events (not at screening), viral load, quality of life and sleep quality will occur at screening and days 1, 28, 90, and 180. Cognitive function will be tested at screening, baseline and day 180.

Primary Endpoint:

* Steady state plasma concentrations of dolutegravir when administered to HIV-infected individuals over the age of 60/65 years.

Secondary Endpoints:

* Safety, tolerability, maintenance of HIV viral load control, quality of life and sleep quality with abacavir/lamivudine/dolutegravir once daily in HIV-infected subjects of 60 years or greater
* Measurement of the metabolic profile in patients over the age of 60 with HIV infection who switch antiretroviral regime (metabonomics)
* Cerebral function via cognitive testing before and after a switch in antiretroviral therapy to dolutegravir containing regimens
* Relationship between genetic polymorphisms and exposure to dolutegravir.

ELIGIBILITY:
Inclusion Criteria:

1. HIV-1 infected males or females
2. Has voluntarily signed informed consent after having enough time to consider the study information.
3. Is willing to comply with the protocol requirements
4. Documentation that the subject is negative for the HLA-B*5701 allele, either on historical sample or if none available, at screening.
5. Aged 60 years and over (approximately 70% of the study participants will be ≥65 year of age), willing to switch therapy as per study protocol with no previous use of dolutegravir
6. Plasma HIV RNA < 50 copies/mL at screening (single re-test allowed) and on at least one other occasion over the last 6-8 months
7. Has a CD4 cell count at screening >50 cells/mm3
8. Currently receiving a stable antiretroviral regimen with no antiretroviral drug switches for at least 3 months prior to planned study baseline.
9. No previous clinically-significant resistance documented on HIV-1 genotypic resistance to NRTIs and INIs
10. Subjects in good health upon medical history, physical exam, and laboratory testing and with a clinically managed cardiovascular disease in the opinion of the Investigator
11. Body mass over 40 kg and body mass index (BMI) above or equal to 18 and below 35
12. Male subjects who are heterosexually active must be willing to use appropriate and consistent dual method contraception during heterosexual intercourse with women of child bearing potential, from screening through to one month post completion of the study. The following combined contraceptive methods are acceptable (please see appendix 3):

    1. Double barrier method:

       * Male Condom combined with a Female Diaphragm with or without a vaginal spermicide* (foam, gel, film, cream, or suppository)
       * Male Condom combined with a Cervical cap** (with spermicide)
    2. Male Condom + one of the following:

       * Combined Oral Contraceptive Pill
       * Combined Contraceptive Patch
       * Combined Vaginal Ring
       * The Progesterone Only Pill
       * Intra-uterine Device (Copper IUD or the IUS)
       * Injectable progestogen (Depo provera®)
       * The progestogen-only Subdermal Implant

Footnotes:

1. *Cervical caps in women who have given birth is less effective than other methods of contraception.
2. **Spermicide should be used with caution as this can potentially increase the rate of HIV-1 transmission.
3. ***It is advised not to use a male and female condom together due to risk of breakage or damage caused by latex friction.

If a female partner has had a total hysterectomy (surgical removal of the womb) or bilateral tubal ligation/clip (surgical sterilization), then she cannot get pregnant and the above section does not apply. If the male subject has had a vasectomy at least 1 month prior to starting the study, he does not need to use any other birth control.

Exclusion Criteria:

1. History or presence of allergy to the study drugs or their components
2. Infected with HIV-2
3. Using any concomitant therapy disallowed as per SPC for the study drugs. The SPC of a drug is updated regularly. The most recent version can be found on http://www.medicines.org.uk/emc/
4. Known acute viral hepatitis including, but not limited to, A, B, or C
5. Known chronic hepatitis B and/or C
6. Tests newly positive for active Hepatitis B (HBsAg positive), or active Hepatitis C (PCR positive) at screening visit
7. Any investigational drug within 30 days prior to the trial drug administration
8. Alanine aminotransferase (ALT) ≥5 times the upper limit of normal (ULN), OR ALT ≥3xULN and bilirubin ≥1.5xULN (with >35% direct bilirubin)
9. Subjects with moderate to severe hepatic impairment (Class B or greater) as determined by Child-Pugh classification
10. Moderate or severe renal impairment (creatinine clearance < 50ml/min)
11. Screening blood result with any grade 3/4 toxicity according to Division of AIDS (DAIDS) grading scale, except: asymptomatic grade 3 glucose, amylase or lipid elevation or asymptomatic grade 4 triglyceride elevation (re-test allowed).
12. Any condition (including drug/alcohol abuse) or laboratory results which, in the investigator's opinion, interfere with the assessments or completion of the trial.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2015-08-04 (Actual); Primary Completion 2017-02-13 (Actual); Study Completion 2017-07-24 (Actual)

PRIMARY OUTCOMES:
Steady state plasma concentrations of dolutegravir when administered to HIV-infected individuals over the age of 60/65 years. | Day 28

SECONDARY OUTCOMES:
Safety on abacavir/lamivudine/dolutegravir once daily in HIV-infected subjects of 60 years or greater - measured by Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events. | Up to day 190
Tolerability on abacavir/lamivudine/dolutegravir once daily in HIV-infected subjects of 60 years or greater- measured by Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events. | Up to day 190
Maintenance of HIV viral load control on abacavir/lamivudine/dolutegravir once daily in HIV-infected subjects of 60 years or greater. | Up to day 190
Quality of life on abacavir/lamivudine/dolutegravir once daily in HIV-infected subjects of 60 years or greater.- Measured by questionnaire | Up to day 190
Sleep Quality on abacavir/lamivudine/dolutegravir once daily in HIV-infected subjects of 60 years or greater - Measured by questionnaire | Up to day 190
Measurement of the metabolic profile in patients over the age of 60 with HIV infection who switch antiretroviral regime (metabonomics) | Up to day 180
Cerebral function via cognitive testing before and after a switch in antiretroviral therapy to a dolutegravir containing regimen | Up to day 180
Relationship between genetic polymorphisms and exposure to dolutegravir as measured by Peak plasma concentration (Cmax) | Day 1
  The results of genetic polymorphisms testing indicating the presence or absence of certain polymorphisms coding for enzymes and transporters responsible for the metabolism of dolutegravir will be correlated with the PK parameter Peak plasma concentration (Cmax). This, for instance, can tell us if the presence of certain alleles makes an individual more likely to metabolise or clear dolutegravir faster or slower.
Relationship between genetic polymorphisms and exposure to dolutegravir as measured by trough concentration (Ctrough) | Day 1
  The results of genetic polymorphisms testing indicating the presence or absence of certain polymorphisms coding for enzymes and transporters responsible for the metabolism of dolutegravir will be correlated with the PK parameter trough concentration (Ctrough). This, for instance, can tell us if the presence of certain alleles makes an individual more likely to metabolise or clear dolutegravir faster or slower.
Relationship between genetic polymorphisms and exposure to dolutegravir as measured by Area under the plasma concentration versus time curve (AUC) | Day 1
  The results of genetic polymorphisms testing indicating the presence or absence of certain polymorphisms coding for enzymes and transporters responsible for the metabolism of dolutegravir will be correlated with the PK parameter Area under the plasma concentration versus time curve (AUC). This, for instance, can tell us if the presence of certain alleles makes an individual more likely to metabolise or clear dolutegravir faster or slower.

CONTACTS AND LOCATIONS:
Overall Officials: Marta Boffito, Principal Investigator — St Stephen's AIDS Trust
Locations (1):
- St Stephen's Centre, Chelsea & Westminster Hospital, London, United Kingdom